CLINICAL TRIAL: NCT06019299
Title: Cluster-randomized Controlled Trial Examining the Effectiveness of Mindfulness-Based Cognitive Therapy for Anxiety and Stress Reduction Within College Students
Brief Title: Cluster-randomized Controlled Trial of Mindfulness-Based Cognitive Therapy Effects on Anxiety and Stress
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Responsible Party: Principal Investigator, Matthew B. Pontifex, Ph.D., Professor of Kinesiology and Psychology, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00008121
Record Dates: First submitted 2023-07-18; First posted 2023-08-31 (Actual); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Anxiety; Stress
Keywords: Mindfulness-Based Cognitive Therapy
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Cluster randomized allocation to Mindfulness-Based Cognitive Therapy intervention or positive control intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive Control (Active Comparator): The control experimental group received training on the utilization of mindfulness-based stress reduction breathing techniques. Participants were instructed to set a timer for 5 minutes in order to engage in mindfulness breathing. Comprehensive instructions were provided during the initial laboratory time, elucidating the method by which participants were to direct their attention towards their breath. Moreover, participants were encouraged to cultivate a non-judgmental attitude when confronted with potential distractions and to subsequently redirect their focus back to their breathing. Participants were advised to integrate this technique into their daily lives as a means to alleviate anxiety and stress.
  Interventions: Behavioral: Mindfulness Practice
- Mindfulness-Based Cognitive Therapy intervention (Experimental): The active experimental group received a mindfulness based cognitive therapy through the Sanvello smartphone application. Participants were encouraged to practice mindfulness daily through the application program "Braving Anxiety," which consisted of 35 modules. The anxiety management program consists of 1) Watch, 2) Read, 3) Listen, 4) Plan, 5) Listen - Mindfulness practice.
  Interventions: Behavioral: Mindfulness Practice

INTERVENTIONS:
Behavioral: Mindfulness Practice — Participants were instructed to practice mindfulness daily using their instructed approaches for a period of 4 weeks.

SUMMARY:
To understand the potential effectiveness of a 4 week Mindfulness-Based Cognitive Therapy intervention delivered using a smartphone application for reducing anxiety and stress within college students.

DETAILED DESCRIPTION:
The objective of this project is to understand the potential effectiveness of a 4 week Mindfulness-Based Cognitive Therapy intervention delivered using a smartphone application for reducing anxiety and stress within college students. Although in-person mindfulness-based cognitive therapy approaches have been found effective for reducing anxiety and stress; given the pervasiveness of anxiety and stress in this population, there is a need to provide alternative and accessible interventions to improve students' mental health. One such approach may be by leveraging existing tools such Sanvello - a free mindfulness-based cognitive therapy smartphone application - which could more easily be deployed across a broader population. Accordingly, using a cluster-randomized controlled design, this intervention will assess the extent to which 4-weeks of using the Sanvello application was effective for reducing anxiety and stress within college students.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in course

Exclusion Criteria:

* Complete inattendance in course during the pretest and study period.
* Opted out of data being available for research use

Ages: 17 Years to 42 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 289 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-04-26 (Actual); Study Completion 2023-04-26 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory | Change from baseline, 4 weeks.
  Trait scale of the Spielberger State-Trait Inventory as an index of trait anxiety
Perceived Stress Scale | Change from baseline, 4 weeks.
  The Perceived Stress Scale-4 as an index of perceived chronic stress levels

CONTACTS AND LOCATIONS:
Overall Officials: Matthew B Pontifex, PhD, Principal Investigator — Michigan State University
Locations (1):
- Department of Kinesiology, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Data sharing will be by request and approval of the Michigan State University Human Research Protections Program with the provision of a data-safety and sharing agreement. No individually identifiable information will be shared.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be available following primary publication of the results.
Access Criteria: By request and completion of an institutional data-safety and sharing agreement.

REFERENCES:
- [Derived] Ellison OK, Bullard LE, Lee GK, Vazou S, Pfeiffer KA, Baez SE, Pontifex MB. Examining efficacy and potential mechanisms of mindfulness-based cognitive therapy for anxiety and stress reduction among college students in a cluster-randomized controlled trial. Int J Clin Health Psychol. 2024 Oct-Dec;24(4):100514. doi: 10.1016/j.ijchp.2024.100514. Epub 2024 Oct 29. PMID 39525940

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/99/NCT06019299/Prot_SAP_000.pdf